CLINICAL TRIAL: NCT01028352
Title: UMCC 2008.62: Prospective Pilot Study Evaluating the Use of Duloxetine for Treatment of Aromatase Inhibitor-associated Musculoskeletal Symptoms in Breast Cancer Patients
Brief Title: Study to Assess Effect of 8 Wks of Duloxetine Therapy on Breast Cancer Patients With Aromatase-Inhibitor Associated Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Lynn Henry, Assistant Professor of Internal Medicine, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2008.062; HUM00022455 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duloxetine (Other)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Patients will be treated with open-label duloxetine:
  * 30 mg daily x 7 days, then
  * 60 mg daily x 3 weeks, then
  * If a patient believes she has experienced a sufficient reduction in pain after 4 weeks of therapy, she will continue taking 60 mg daily for weeks 5-8
  * If a patient does not believe she has experienced a sufficient reduction in pain after 4 weeks of therapy, she will have the option of increasing the dose to 60 mg twice daily for weeks 5-8.
  * After completion of 8 weeks of therapy, patients who wish to discontinue therapy will taper off the drug over 1 week (50% decrease for 4 days, then additional 50% decrease for 3 days). Patients may continue therapy off-study at the discretion of their treating physician.
  Other Names: Cymbalta

SUMMARY:
Many women with breast cancer who are treated with aromatase inhibitor medications develop aches and pains during treatment, and some develop numbness and tingling in their hands and feet. Some examples of aromatase inhibitor medications include anastrozole (Arimidex), exemestane (Aromasin), and letrozole (Femara). Frequently, pain medications do not work very well to relieve the pain. Duloxetine (Cymbalta) is a medication that was originally developed to treat depression. It has also been found to relieve pain that occurs in people with diabetes, fibromyalgia, arthritis, and other painful conditions. In this study we are testing to see if duloxetine will help treat the pain that can occur in women treated with aromatase inhibitors.

DETAILED DESCRIPTION:
Aromatase inhibitor (AI) therapy is commonly used for treatment of postmenopausal women with hormone receptor-positive breast cancer. The most common toxicities are arthralgias and myalgias, which can be difficult to manage and necessitate discontinuation of therapy in up to 10% of patients. One potential interventional approach is with a pharmaceutical agent such as duloxetine, which has been shown to be effective for treatment of other types of chronic pain, including fibromyalgia and diabetic neuropathic pain.

The primary objective of this pilot study is to determine the proportion of breast cancer patients with AI-associated musculoskeletal symptoms who experience a 30% reduction in average pain score from baseline to 8 weeks due to duloxetine treatment. Participants will be treated with duloxetine for 8 weeks. Questionnaires to evaluate pain, functional status, depression, menopausal symptoms, and sleep difficulties will be administered at baseline and after 2, 4, 6, and 8 weeks of therapy. In addition, 10 milliliters blood of will be drawn from the subjects at baseline for future pharmacogenetic evaluation. If the results of this pilot study suggest that the efficacy of duloxetine therapy is greater than that expected from placebo based on historical controls, then these data will be used to design future prospective, placebo-controlled, randomized trials of treatment with duloxetine in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Histologically proven stage 0-III invasive carcinoma of the breast that is ER and/or PR positive by immunohistochemical staining, who are receiving a standard dose of aromatase inhibitor (AI) therapy (letrozole 2.5mg once daily or exemestane 25mg once daily or anastrozole 1mg once daily). Women with oligometastatic disease may be included at the discretion of the principal investigator. Surgical resection, chemotherapy, and radiation therapy must have been completed at the time of study enrollment, with the exception of trastuzumab;
* AI therapy has been ongoing for ≥ 2 weeks and treatment is expected to continue;
* AI-associated musculoskeletal symptoms, defined as:

  * Grade 1 or higher musculoskeletal pain that developed or worsened (6 or 7 on CGICS) during AI therapy or
  * Grade 1 or higher sensory neuropathy that developed or worsened (6 or 7 on CGICS) during AI therapy;
* Average pain of ≥4 on the 11-point Likert scale of question #5 of the Brief Pain Inventory;
* ECOG performance status 0-2;
* Willing and able to sign an informed consent document.

Exclusion Criteria:

* Known hypersensitivity to duloxetine or any of the inactive ingredients;
* New musculoskeletal pain that is due specifically to fracture or traumatic injury;
* Treatment with monoamine oxidase inhibitors (MAO-I) within 14 days of enrollment;
* Concurrent treatment with phenothiazines (including thioridazine), propafenone, flecainide, triptans, MAO-Is, SSRIs, SNRIs, or tricyclic antidepressants;
* Currently primary psychiatric diagnosis (schizophrenia, psychosis) or suicidal ideation, history of bipolar disorder, or seizure disorder;
* Chronic liver disease, end stage renal disease, or creatinine clearance < 30 mL/min as defined by the Cockroft-Gault equation;
* Uncontrolled narrow-angle glaucoma or clinically significant coagulation disorder;
* Pregnant or breast feeding;
* History of alcohol or other substance abuse or dependence within the year prior to enrollment;
* Serious or unstable medical condition that could likely lead to hospitalization during the course of the study or compromise study participation.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Henry NL, Banerjee M, Wicha M, Van Poznak C, Smerage JB, Schott AF, Griggs JJ, Hayes DF. Pilot study of duloxetine for treatment of aromatase inhibitor-associated musculoskeletal symptoms. Cancer. 2011 Dec 15;117(24):5469-75. doi: 10.1002/cncr.26230. Epub 2011 Jun 20. PMID 21692065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2008 and May 2010 35 subjects enrolled and completed baseline questionnaires in the University of Michigan comprehensive cancer center's outpatient hematolgy / oncology clinic
Groups:
- Duloxetine: Participants took 30 mg oral capsules once a day for 7 days, then 60 mg per mouth once per day for 21 days. After 4 weeks if pain had decreased, subjects continued 60 mg. per mouth once per day for 4 weeks. If pain had not decreased, subjects took 60 mg twice per day per mouth for 4 weeks. 5 Questionnaires were administered at baseline and every 2 weeks for 8 weeks; medication was tapered at the end of study.
Period: Overall Study
Arm/Group | Duloxetine
Started | 35
Completed | 29
Not Completed | 6
Not completed — Ineligible due to baseline average pain | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Experience 30% Reduction in Average Pain Score From Baseline to 8 Weeks Due to Duloxetine Therapy.
Description: Subjects were considered evaluable if they met all eligibility criteria and took at least one dose of duloxetine. Average pain was measured using Wisconsin Brief Pain Inventory Questionnaire.(BPI) The BPI is a 17-item patient self-rating scale that assessed sensory & reactive components of pain. The BPI uses 0 to 10 numeric rating scales for item rating.Since pain can be variable,the BPI asks patients to rate pain at completing questionnaire, and also at its worst, least, and average over the previous 24 hours. The primary endpoint is based on the 24-hour avg pain as reported on BPI.
Time Frame: 8 weeks
Population: Subjects were considered evaluable for the primary endpoint if they met all eligibility criteria and took at least one dose of duloxetine
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
percentage of participants | 72.4

2. Secondary Outcome: Decrease in Average Pain With 8 Weeks of Duloxetine Therapy. (Sustained)
Description: A secondary measure is the percentage of patients treated with duloxetine who experience a sustained 30% reduction in average pain score from baseline to 8 weeks. Sustained 30% reduction is defined as at least 30% reduction in 24-hour average pain severity at the 8 week endpoint, with a 30% reduction from baseline at a visit at least 2 weeks prior to the last visit, and at least 20% reduction from baseline at every visit in between.
Time Frame: Baseline, 2, 4 , 6 and 8 weeks
Measure: Number (95% Confidence Interval); unit: %of participants with 30% pain reduction
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
%of participants with 30% pain reduction | 60.9 [48.6 to 73.1]

ADVERSE EVENTS:
Time Frame: 1 year and 5 months
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 7/29
OTHER ADVERSE EVENTS (reported when occurring in more than 2.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=29)
Fatigue (General disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 6 (6)
Headache (General disorders) | 5 (5)
Dry mouth (General disorders) | 5 (5)
Drowsiness (General disorders) | 4 (4)
Heartburn (Gastrointestinal disorders) | 3 (3)
Anxiety (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No